CLINICAL TRIAL: NCT00833118
Title: Tongue Pull Versus Jaw Thrust
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sorin Brull, M.D., Mayo Clinic Florida
Other Study IDs: 07-004837
Record Dates: First submitted 2009-01-29; First posted 2009-01-30 (Estimated); Last update posted 2010-02-12 (Estimated); Status verified 2010-02

CONDITIONS: Surgery
Keywords: Surgery; General Anesthesia; Intubation
MeSH Terms: interventions — Intubation

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (1):
- Intubation
  Interventions: Procedure: Jaw thrust maneuver (Intubation)

INTERVENTIONS:
Procedure: Jaw thrust maneuver (Intubation) — Visualization of Larygnoscopic anatomy during intubation

SUMMARY:
This protocol seeks to determine the efficacy and reliability of a simple maneuver, the jaw thrust maneuver, in addition to cricoid pressure, in improving visualization of airway anatomy during video laryngoscopy. Hypothesis: The grade of view of the glottis as determined by the modified Cormack and Lehane grading system in anesthetized patients will improve by performing a jaw thrust maneuver during video laryngoscopy with compared with video laryngoscopy alone. Similarly, the grade of the view during cricoid pressure will also improve with a jaw thrust maneuver.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18
2. Undergoing surgery and general anesthesia with endotracheal intubation
3. Able to give informed consent

Exclusion Criteria:

1. Trauma patients or emergent cases.
2. Patients who are unable to understand the proposed study
3. Patients who refuse participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male or female scheduled for surgery and undergoing intubation for general anesthesia administration
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2008-11; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sorin Brull, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Florida, Jacksonville, Florida, United States